CLINICAL TRIAL: NCT01643395
Title: VertebrOpLasty Versus Conservative Treatment in Acute Non Osteoporotic Vertebral Fractures
Acronym: VOLCANO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0122
Record Dates: First submitted 2012-07-13; First posted 2012-07-18 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Vertebral Compression Fracture; Spinal Trauma
Keywords: Trauma; vertebral; compression fracture; spinal; acute; vertebroplasty; conservative treatment
MeSH Terms: conditions — Wounds and Injuries; Fractures, Compression | interventions — Vertebroplasty; Conservative Treatment

ARMS (2):
- vertebroplasty (Experimental)
  Interventions: Other: vertebroplasty
- conservative therapy (brace) (Other)
  Interventions: Other: conservative therapy

INTERVENTIONS:
Other: vertebroplasty — Vertebroplasty consists in the injection of cement (PMMA) in the damaged vertebral body to prevent further collapse
  Arms: vertebroplasty
Other: conservative therapy — The study is a prospective, randomized trial comparing conservative treatment (brace) and vertebroplasty in acute (less than 15 days after trauma) traumatic vertebral compression fracture (VCF) type A according Magerl classification.
  Arms: conservative therapy (brace)

SUMMARY:
The purpose of this protocol is to prove the efficacy of vertebroplasty in patients suffering from acute non osteoporotic vertebral compression fracture.

Vertebroplasty consists in the injection of cement (PMMA) in the damaged vertebral body to prevent further collapse.

Our study will compare vertebroplasty versus conservative therapy (brace).

DETAILED DESCRIPTION:
The study is a prospective, randomized trial comparing conservative treatment (brace) and vertebroplasty in acute (less than 15 days after trauma) traumatic vertebral compression fracture (VCF) type A according Magerl classification

ELIGIBILITY:
Inclusion Criteria:

* 18 - 70 year old
* volunteers
* Vertebral compression fractures Magerl type A
* Acute Trauma (less than 15 days)
* Between T5 and L5
* Patient able to undergo both vertebroplasty and conservative treatment
* Consent form obtained

Exclusion Criteria:

* Neural arch fracture
* C1 to T4 fracture
* Neurologic symptoms caused by the fracture
* Encephalic trauma with Glasgow Coma Scale less than 15
* Ongoing cancer
* Routine painkillers intake
* Local or systemic infection
* Coagulation's disorder
* Pregnancy
* Involvement in an another clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Disability scale | at 1 month

SECONDARY OUTCOMES:
Spine radiological measurements | at 1, 3 and 6 months
Disability and qol | at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel CHABERT, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Chabert E, Hugonnet E, Kastler A, Sakka L, Rabbo FA, Zerroug A, Coudeyre E, Pereira B, Coll G. Vertebroplasty versus bracing in acute vertebral compression fractures: A prospective randomized trial. Ann Phys Rehabil Med. 2023 Sep;66(6):101746. doi: 10.1016/j.rehab.2023.101746. Epub 2023 Apr 6. PMID 37030247